CLINICAL TRIAL: NCT00345605
Title: A Randomized, Double-Blind, Crossover Study of Sodium Phenylbutyrate and Low-Dose Arginine Compared to High-Dose Arginine Alone on Liver Function, Ureagenesis and Subsequent Nitric Oxide Production in Patients With Argininosuccinic Aciduria
Brief Title: Arginine and Buphenyl in Patients With Argininosuccinic Aciduria (ASA), a Urea Cycle Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brendan Lee (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); Rare Diseases Clinical Research Network (Network); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Brendan Lee, MD, PhD, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RDCRN 5102; U54HD061221 (NIH)
Record Dates: First submitted 2006-06-26; First posted 2006-06-28 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2015-10

CONDITIONS: Argininosuccinic Aciduria; Amino Acid Metabolism, Inborn Errors; Urea Cycle Disorders
Keywords: Argininosuccinic Acid Lyase Deficiency; ASA
MeSH Terms: conditions — Argininosuccinic Aciduria; Amino Acid Metabolism, Inborn Errors; Urea Cycle Disorders, Inborn | interventions — 4-phenylbutyric acid; Arginine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HDA (Experimental): High Dose Arm
  Wash-out then 7 days of:
  Arg 500 mg/kg/d or 10 g/m2 BSA Placebo instead of NaPBA
  Interventions: Drug: Sodium Phenylbutyrate; Drug: Arginine
- LDA (Experimental): Low Dose Arm
  Wash-out followed by 7 days of:
  Arg 100 mg/kg/d or 2 g/m2 BSA NaPBA 500 mg/kg/d or 10 g/m2 BSA
  Interventions: Drug: Sodium Phenylbutyrate; Drug: Arginine

INTERVENTIONS:
Drug: Sodium Phenylbutyrate — None will be administered during the washout period; 500 mg/kg/day or 10 grams/m2 will be administered during the first one week treatment period in addition to arginine
  Other Names: Buphenyl-TM
Drug: Arginine — Standard therapeutic dose of 500 mg/kg/day or 10 grams/2 will be administered during the washout periods, during the first one week treatment period when receiving arginine plus Buphenyl, 100 mg/kg/day or 2 grams/m2 will be administered, during the second treatment week, when receiving arginine alone, 500 mg/kg/day or 10 grams/m2 will be administered

SUMMARY:
Urea cycle disorders are inherited illnesses in which the body does not produce enough of the chemicals that remove ammonia, a byproduct of protein metabolism, from the blood stream. Elevated ammonia levels can lead to brain damage and death. Argininosuccinic aciduria (ASA) is a type of urea cycle disorder that is characterized specifically by high levels of argininosuccinic acid, a chemical involved in the urea cycle. People with ASA are at risk for serious liver damage, which may be due to the elevated levels of argininosuccinic acid. Sodium phenylbutyrate (Buphenyl-TM) is a drug that has been used to treat other types of urea cycle disorders. This study will evaluate whether Buphenyl-TM in conjunction with decreased arginine dose (in addition to a normal regimen of protein) will improve short-term liver function and decrease plasma citrulline and ASA levels in people with ASA.

DETAILED DESCRIPTION:
The cause of liver damage in people with ASA is unknown. However, because ASA is the only urea cycle disorder that is characterized by both liver damage and elevated levels of argininosuccinic acid, researchers believe that the elevated acid levels cause the liver damage. Common treatments for urea cycle disorders include a low-protein diet and arginine supplementation, which, when combined, help to decrease ammonia levels in the blood. Buphenyl-TM may aid in lowering ammonia and argininosuccinic acid levels. Although Buphenyl-TM has been FDA-approved for use in people with some types of urea cycle disorders, there is little information on the effectiveness of the drug in children with ASA. This study will evaluate whether treatment of ASA patients with Buphenyl-TM in conjunction with lowered doses of arginine improves liver function as measured by short-term assessment of synthetic activity and the use of stable isotope tracers to assess ureagenesis and nitric oxide production.

Initially, participants in this double-blind, placebo-controlled, crossover study will undergo a 3-day washout period during which no Buphenyl-TM will be given. They will then be randomly assigned to one of two groups: either Buphenyl-TM (500 mg/kg/day or 10 grams/m2) and arginine (100 mg/kg/day or 2 grams/m2)), or arginine alone (500 mg/kg/day or 10 grams/m2). Participants will remain on this initial treatment arm for 1 week, at the conclusion of which an assessment of hepatic synthetic function, ureagenesis, and nitric oxide production will be performed. After this assessment, participants will undergo a second 3-day washout and then crossover to the other treatment arm for 1 week. At the end of the 1-week treatment period, a second assessment will be performed. During the washout period before each treatment period, no Buphenyl-TM will be administered, and arginine will be administered at the standard therapeutic dose of 500 mg/kg/day or 10 grams/2.

ELIGIBILITY:
Inclusion Criteria:

* Has confirmed diagnosis of ASA by amino acid or enzyme assay
* Has a history of adequate compliance to the diet and treatment
* Able to take oral or G-tube medication
* Able to perform 24 hour urine collection
* Agrees to travel to Baylor College of Medicine
* If female, of child bearing potential, and sexually active, agrees to use an acceptable method of birth control
* Greater than 5 years of age

Exclusion Criteria:

* Has a history of congestive heart failure, severe renal insufficiency, or any condition that causes sodium retention or edema
* Currently taking Probenecid, Haloperidol, Valproate or oral corticosteroids
* Pregnant or lactating
* Currently being treated for an acute illness
* Has co-morbid associations causing difficulties in the detection of hyperammonemic episodes, liver damage, or difficulties in the diet compliance
* Has known hypersensitivity to sodium phenylbutyrate
* Has taken any experimental medication within the last 30 days
* Has renal insufficiency with creatinine greater than 1.5 mg/dl at screening

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-02; Primary Completion 2011-05 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Lee, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Annet L, Materne R, Danse E, Jamart J, Horsmans Y, Van Beers BE. Hepatic flow parameters measured with MR imaging and Doppler US: correlations with degree of cirrhosis and portal hypertension. Radiology. 2003 Nov;229(2):409-14. doi: 10.1148/radiol.2292021128. Epub 2003 Sep 11. PMID 12970464
- [Background] Lu LG, Zeng MD, Wan MB, Li CZ, Mao YM, Li JQ, Qiu DK, Cao AP, Ye J, Cai X, Chen CW, Wang JY, Wu SM, Zhu JS, Zhou XQ. Grading and staging of hepatic fibrosis, and its relationship with noninvasive diagnostic parameters. World J Gastroenterol. 2003 Nov;9(11):2574-8. doi: 10.3748/wjg.v9.i11.2574. PMID 14606100
- [Background] Scaglia F, Marini J, Rosenberger J, Henry J, Garlick P, Lee B, Reeds P. Differential utilization of systemic and enteral ammonia for urea synthesis in control subjects and ornithine transcarbamylase deficiency carriers. Am J Clin Nutr. 2003 Oct;78(4):749-55. doi: 10.1093/ajcn/78.4.749. PMID 14522733
- [Background] Lee B, Yu H, Jahoor F, O'Brien W, Beaudet AL, Reeds P. In vivo urea cycle flux distinguishes and correlates with phenotypic severity in disorders of the urea cycle. Proc Natl Acad Sci U S A. 2000 Jul 5;97(14):8021-6. doi: 10.1073/pnas.140082197. PMID 10869432
- [Background] Brusilow SW, Maestri NE. Urea cycle disorders: diagnosis, pathophysiology, and therapy. Adv Pediatr. 1996;43:127-70. No abstract available. PMID 8794176

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 subjects with argininosuccinic aciduria were recruited at Baylor College of Medicine from May 2008 to December 2010.
Pre-assignment Details: patients were randomly assigned to one of the two arms HDA or LDA after treatment and an interval the same patients returned and received the crossover treatment LD or HDA depending.
Groups:
- High Dose First: High dose arm 3 day wash-out followed by 7 days of: Arg 500 mg/kg/d or 10 g/m2 BSA Placebo instead of NaPBA interval then: Arg 100 mg/kg/d or 2 g/m2 BSA NaPBA 500 mg/kg/d or 10 g/m2 BSA
- Low Dose First: low dose arm 3 day wash-out followed by 7 days of: Arg 100 mg/kg/d or 2 g/m2 BSA NaPBA 500 mg/kg/d or 10 g/m2 BSA interval then: Arg 500 mg/kg/d or 10 g/m2 BSA Placebo instead of NaPBA
Period: Initial Washout
Arm/Group | High Dose First | Low Dose First
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Arm 1
Arm/Group | High Dose First | Low Dose First
Started | 6 | 6
Completed | 6 | 5
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Interval
Arm/Group | High Dose First | Low Dose First
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Crossover Wash-out
Arm/Group | High Dose First | Low Dose First
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Arm 2, Opposite Treatment
Arm/Group | High Dose First | Low Dose First
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | High-dose Arginine vs Low-dose Arginine Plus Buphenyl
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Measures of Liver Function: AST and ALT
Description: Plasma aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels were measured.
Time Frame: Measured after each 1-week treatment period
Measure: Mean (Standard Error); unit: IU/L
Groups:
- Low-dose Arginine Plus Buphenyl: Participants will undergo treatments in the following order: a 3-day washout period; a 1-week treatment period of sodium phenylbutyrate (Buphenyl-TM) plus arginine; a 3-day washout period; a 1-week treatment period of arginine alone.
- High Dose Arginine Alone: Participants will undergo treatments in the following order: a 3-day washout period; a 1-week treatment period of arginine alone; a 3-day washout period; a 1-week treatment period of sodium phenylbutyrate (Buphenyl-TM) plus arginine
Arm/Group | Low-dose Arginine Plus Buphenyl | High Dose Arginine Alone
Number analyzed (Participants) | 11 | 11
IU/L
  Plasma AST | 36.2 (10.9) | 52 (15.7)
  ALT | 31.7 (9.55) | 57.86 (17.44)
Statistical Analysis 1: Comparison: Low-dose Arginine Plus Buphenyl vs High Dose Arginine Alone; For sample size calculation, we used the means and standard deviation for PT, PTT. Assuming r=0.5 between two measurements from the same subject, 12 subjects would provide a power of 0.8 to detect a 10% reduction in primary endpoints at an alpha value of 0.05; Test type: Superiority or Other; Slope = 0.5 — Assuming r=0.5 between two measurements from the same subject, 12 subjects would provide a power of 0.8 to detect a 10% reduction in primary endpoints at an alpha value of 0.05

2. Secondary Outcome: Argininosuccinic Acid Levels
Time Frame: Measured after each 1-week treatment period
Measure: Median (Inter-Quartile Range); unit: micromole/l
Arm/Group | High-dose Arginine Alone | Low-dose Arginine Plus Buphenyl
Number analyzed (Participants) | 11 | 11
micromole/l | 69 [44 to 165] | 53 [29 to 118]

3. Secondary Outcome: Arginine Levels
Time Frame: Measured after each 1-week treatment period
Measure: Median (Inter-Quartile Range); unit: micromoles/L
Arm/Group | High-dose Arginine Alone | Low-dose Arginine Plus Buphenyl
Number analyzed (Participants) | 11 | 11
micromoles/L | 129 [83 to 197] | 53 [41 to 61]

4. Secondary Outcome: Urea Production Rate
Time Frame: Measured after each 1-week treatment period
Measure: Mean (Standard Deviation); unit: micromoles/kg/hr
Arm/Group | High-dose Arginine Alone | Low-dose Arginine Plus Buphenyl
Number analyzed (Participants) | 11 | 11
micromoles/kg/hr | 215 (56) | 97 (35)

5. Primary Outcome: Measures of Liver Function: PT and PTT
Description: Prothrombin time (PT) and partial thromboplastin time (PTT) were measured PT measures factors I (fibrinogen), II (prothrombin), V, VII, and X, while PTT is a performance indicator of the efficacy of the common coagulation pathways.
Time Frame: Measured after each 1-week treatment period
Measure: Mean (Inter-Quartile Range); unit: seconds
Arm/Group | Low-dose Arginine Plus Buphenyl | High Dose Arginine Alone
Number analyzed (Participants) | 11 | 11
seconds
  PT | 14.25 [13.7 to 14.6] | 13.8 [13.6 to 14.37]
  PTT | 30.91 [29.55 to 32.54] | 30.98 [29.16 to 31.74]

6. Primary Outcome: Measures of Liver Function: Coagulation Factors
Description: Plasma levels of coagulation factors I and IX were used as measures of hepatic synthetic function since the treatment duration was short.
Time Frame: Measured after each 1-week treatment period
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Low-dose Arginine Plus Buphenyl | High Dose Arginine Alone
Number analyzed (Participants) | 11 | 11
mg/dL
  I | 222.22 (47.26) | 229.77 (62.96)
  IX | 105.33 (33.2) | 98.36 (21.03)

7. Primary Outcome: Measures of Liver Function: INR
Description: The result (in seconds) for a prothrombin time performed on a normal individual will vary according to the type of analytical system employed. This is due to the variations between different batches of manufacturer's tissue factor used in the reagent to perform the test. The INR was devised to standardize the results. Each manufacturer assigns an ISI value (International Sensitivity Index) for any tissue factor they manufacture. The ISI value indicates how a particular batch of tissue factor compares to an international reference tissue factor. The ISI is usually between 1.0 and 2.0. The INR is the ratio of a patient's prothrombin time to a normal (control) sample, raised to the power of the ISI value for the analytical system being used.
Time Frame: Measured after each 1-week treatment period
Measure: Mean (Inter-Quartile Range); unit: seconds
Arm/Group | Low-dose Arginine Plus Buphenyl | High Dose Arginine Alone
Number analyzed (Participants) | 11 | 11
seconds | 14.2 [13.7 to 14.6] | 13.8 [13.6 to 14.3]

ADVERSE EVENTS:
Time Frame: during both of the 7 day treatment phases
Arm/Group | High-dose Arginine Alone | Low-dose Arginine Plus Buphenyl
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-dose Arginine Alone (N=12) | Low-dose Arginine Plus Buphenyl (N=12)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hyperammonemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No